CLINICAL TRIAL: NCT03143881
Title: Assessment Of Patient Knowledge And Effects Of Educational Strategies In Un- And Under-Insured Heart Failure Patients Presenting To The Emergency Department For Care
Brief Title: Assessment Of Educational Strategies In Heart Failure Patients Presenting To The Emergency Department For Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Vishwaratn Asthana, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32676
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention patients will receive personalized education regarding their condition, pre- and post-testing of their HF knowledge base, and ED standard of care during the enrollment (index) visit. Patients will then be contacted via telephone 30 days post-index visit for re-testing and reinforcement of previously learned material.
  Interventions: Behavioral: Education
- Control (No Intervention): Control patients will receive ED standard of care.

INTERVENTIONS:
Behavioral: Education — Standardized information on the etiology of HF, mechanisms and side effects of medications prescribed, strategies for minimizing exacerbations, and warning signs of worsening clinical status will be discussed with the patient.
  Arms: Intervention

SUMMARY:
This study evaluates the impact of a new education-based intervention on outcomes in un- and under-insured Heart Failure (HF) patients presenting to the Emergency Department (ED) for care. Intervention patients will receive personalized education regarding their condition, pre- and post-testing of their HF knowledge base, and ED standard of care during the enrollment (index) visit. Patients will then be contacted via telephone 30 days post-index visit for re-testing and reinforcement of previously learned material. Patients in the control group will receive ED standard of care.

DETAILED DESCRIPTION:
In 2015, 12.8% of adults ages 19-64 in the United States lacked any form of health insurance. An even greater number fell under the umbrella of under-insured. Studies indicate that the un- and under-insured receive less preventive care, are diagnosed at more advanced disease stages, and have higher mortality rates than their insured counterparts, due to the lack of accessible primary care services. These issues are most readily evident in patients with chronic conditions. When a preventable, chronic condition worsens, these patients have no choice but to visit the ED to address their most immediate health concerns, leaving the underlying chronic problem untreated. HF is a particularly burdensome chronic problem for patients of all socioeconomic statuses and one of the leading causes of ED and hospital readmissions.

Numerous educational efforts have been tested in an attempt to reduce HF readmissions but have met with mixed results. Consequently, HF patients are generally seen as refractory to educational and management strategies. The investigators propose here a new, targeted educational intervention designed to improve patient outcomes and readmission rates in un- and underinsured HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-existing documented diagnosis of HF presenting to the ED

Exclusion Criteria:

* 1) Patients in unstable condition requiring immediate medical attention, 2) hemodynamically unstable, 3) age < 18 years, and/or 4) incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in ED revisits | 30 and 90 days
  Change in the number of HF-specific ED revisits over the 30- and 90-day periods, pre- and post-index visit.
Change in hospital readmissions | 30 and 90 days
  Change in the number of HF-specific hospital readmissions over the 30- and 90-day periods, pre- and post-index visit.

SECONDARY OUTCOMES:
Days alive and out of hospital (DAOH) | 365 days (1 year)
  Days alive and out of hospital (DAOH) over a 365 day period post-index visit

CONTACTS AND LOCATIONS:
Overall Officials: Vishwaratn Asthana, Principal Investigator — Baylor College of Medicine; William Peacock, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: Undecided